CLINICAL TRIAL: NCT01162057
Title: The Effect of Hemodialysis on Hearing in Hemodialysis Patients
Brief Title: The Effect of Hemodialysis on Hearing
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: N. Berar-Yanay, MD, Nephrology Institute, Hillel Yaffe Medical Center
Other Study IDs: 42-2008
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: Hearing
Keywords: Hemodialysis; Hearing; Hemodialysis patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The inner ear contains transporters that are responsible for maintaining a strict homeostatic environment, necessary for transmission and transduction of sound waves. Hemodialysis affects the body's composition including the aspects regulated by these transporters (pH, osmolarity, Na, K). We wish to observe if hemodialysis affects hearing, and if so, by which parameters.

ELIGIBILITY:
Inclusion Criteria:

* patients on hemodialysis

Exclusion Criteria:

* known hearing defect

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing regular thrice-weekly hemodyalysis
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-08